CLINICAL TRIAL: NCT00897780
Title: Combined Biofeedback With Virtual Reality in the Treatment of Pediatric Headache
Acronym: VR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Itai Berger, MD, HAdassah-Hebrew University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HMO-0445-08
Record Dates: First submitted 2009-05-10; First posted 2009-05-12 (Estimated); Last update posted 2009-05-12 (Estimated); Status verified 2009-05

CONDITIONS: Chronic Headache
Keywords: Headache; Pediatric; Virtual Reality; Biofeedback
MeSH Terms: conditions — Headache Disorders; Headache | interventions — Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Biofeedback with virtual reality — Participant will use biofeedback technique in combination with virtual reality technique
  Other Names: VR; Biofeedback

SUMMARY:
The objective of the study is to examine the effect of combined treatments (biofeedback with virtual reality) for pediatric chronic headache.

DETAILED DESCRIPTION:
Chronic headache is a common symptom in children. Pharmacologic treatment has only a limited productivity and several known adverse reactions. Despite the frequency and chronicity of pediatric headache, validated treatment paradigms are currently inadequate.

Biofeedback is a medical treatment in which physiologic markers like heart rate, breathing rate, EMG, EEG, or electrodermal activity are measured and displayed back to the patient. The patient can then attempt to modulate physiology to achieve a certain feedback goal,such as slowing heart or breath rate, or relaxing certain muscles. Numerous psychophysiologic studies have been conducted that examine the effect of biofeedback alone on physiology as well as various clinical conditions. Clinical trials for chronic headaches have found that biofeedback was more effective in the treatment of headache when compared to pure drug therapy.

A number of recent distraction interventions for acute pain in children and adolescents have employed virtual reality technology in conjunction with either a passive distraction stimulus, such as a movie, or an interactive distraction activity, such as a computer game. However, the actual benefit of VR technology over and above the benefits of the distracting stimulus that is experienced through the VR equipment has not been adequately tested in children.

The objective of this study is to combine virtual reality with biofeedback in order to increase the effectivity of both techniques in decreasing chronic headache frequency and pain degree in the pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* 9-18 years old children suffering from chronic headache diagnosed by pediatric neurologist
* Exclusion of Other disorders causing chronic headache

Exclusion Criteria:

* Children younger than 9 years or olde than 18.
* Children who do not fulfill headache criteria as described in the International Headache Society
* Children who were not examined by a certified pediatric neurologist

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-09 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in headache frequency and pain degree among participants | 6 weeks